CLINICAL TRIAL: NCT04652089
Title: The Effect of Seven-day Simvastatin Administration on Emotional Processing, Reward Processing, and Inflammation in Healthy Volunteers
Brief Title: 7-day Simvastatin and Emotional Processing
Acronym: SSTEP-HV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R69606/RE001
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2020-12

CONDITIONS: Depression; Inflammation
Keywords: Depression; Inflammation
MeSH Terms: conditions — Depression; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Participants will be randomly allocated to one of two groups (simvastatin or placebo) and take the assigned medication for 7 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: Simvastatin (Experimental): Simvastatin 20mg capsule once a day for 7 days
  Interventions: Drug: Simvastatin 20mg
- Control arm: Placebo (Placebo Comparator): Placebo capsule once a day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin 20mg — Simvastatin 20mg once a day for 7 days
  Arms: Experimental arm: Simvastatin
Drug: Placebo — Placebo once a day for 7 days
  Arms: Control arm: Placebo

SUMMARY:
Work in our group has revealed that short-term (7-day) administration of antidepressants produces positive biases in the processing of emotional information in healthy volunteers. Such effect might be an important neuropsychological mechanism of antidepressant action.

The current study will investigate the effect of seven-day administration of simvastatin 20mg on emotional and reward processing tasks in healthy volunteers. There is evidence that statins may exert antidepressant effects via anti-inflammatory and anti-oxidant pathways, and it is therefore predicted that simvastatin will have positive effects on emotional and reward processing.

DETAILED DESCRIPTION:
Depression is common and associated with considerable health disability (Kassebaum-2016). Traditional antidepressants mainly work by modulating monoamine levels in the synaptic cleft (Harmer-2017); however, the evidence that depression is caused by impaired serotonin or noradrenaline activity is weak and inconsistent (Cowen-2015), and indeed current antidepressant strategies remain burdened by partial efficacy, poor side-effects profile, and a slow onset of therapeutic action (Penn-2012). Therefore, there is a pressing need to develop antidepressant medications with novel non-monoaminergic mechanisms of action (Jha-2018) - or, conversely, to identify alternative pathophysiological pathways leading to depression that can be targeted with new drugs. Intriguingly, there is growing evidence that both peripheral and central inflammation play a role in the pathophysiology of depression (Miller-2017).

Patients with depression consistently show negative biases in emotional processing, which are believed to play a key role in the aetiology and maintenance of their clinical symptoms (Roiser-2013). Overall, robust evidence suggests that early changes in emotional processing can serve as valid surrogate markers of antidepressant efficacy (Harmer-2017); for example, seven days' treatment with selective serotonin and noradrenaline reuptake inhibitors (citalopram and reboxetine respectively) compared to placebo decreases the recognition of negative facial expressions and recall of negative versus positive stimuli in healthy volunteers (Harmer-2004). Conversely, another study using the pro-inflammatory cytokine interferon-α showed that inflammatory-mediated depression can be associated with an increased recognition of negative facial expressions (Cooper-2017). Furthermore, depression associated with inflammation is characterised by significant symptoms of anhedonia (Miller-2017), which has been linked to diminished neural responses to reward anticipation (Felger-2017). Such reward-deficit is particularly refractory to conventional serotoninergic and noradrenergic antidepressants (McCabe-201), and even the antidepressant bupropion (a noradrenaline and dopamine reuptake inhibitor), whilst inducing positive changes in emotional processing, appears not to improve reward processing (Walsh-2018). However, the reversal of this deficit in reward processing is still considered as a valuable marker of target engagement for anti-inflammatory drugs in depression, as a more sensitive outcome measure than traditional rating scales designed to capture the global clinical symptomatology (Miller-2017).

The 3-hydroxy-3-methylglutaryl-CoA reductase inhibitors or statins are recommended and have been widely used since the '80s for the primary and secondary prevention of cardiovascular diseases (NICE 2014). It is now established that these medications have significant anti-inflammatory effects that are independent from their lipid-lowering properties (Jain-2005), as well as appearing early in treatment only after seven day of administration (Macin-2011). Statins are considered extremely safe drugs: their more common side-effect are muscle pain or weakness (usually mild and quickly responding to stopping or switching medication) and elevation of liver transaminases (significant only in case of pre-existing hepatic disease), whereas more serious adverse events include rhabdomyolysis (very rare but severe myopathy associated with elevated creatine kinase and myoglobinuria), new-onset diabetes mellitus (in predisposed individual with pre-existing hyperglycaemia), and haemorrhagic stroke (in patients with prior haemorrhagic stroke or lacunar infarct); however, clinical trials have ultimately concluded that such adverse events attributed to statin therapy in routine practice are not actually caused by it (Collins-2016). Other common (≥ 1/100, < 1/10) but usually mild side-effects include: nasopharyngitis, pharyngo-laryngeal pain, epistaxis, headache, and gastrointestinal disturbances (constipation, diarrhoea, flatulence, dyspepsia, nausea). Importantly, a potential antidepressant effect for statins has been confirmed in animals (Kilic-2012), as well as clinically in observational (Parsaik-2014) and interventional studies (Salagre-2016). Although their anti-inflammatory and anti-oxidant properties have been proposed, the precise mechanisms underlying the antidepressant effects of statins remain unclear, therefore further translational studies have been advocated in order to elucidate this aspect (Köhler-Forsberg-2017).

In this exploratory study, we will investigate the effect of seven-day administration of simvastatin 20mg once daily compared to placebo on emotional and reward processing tasks in 50 healthy volunteers. In view of the previous evidence that statins may exert antidepressant effects via anti-inflammatory and anti-oxidant pathways, we predict that simvastatin will have positive effect on emotional and reward processing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-50 years
* Sufficiently fluent English to understand and complete the tasks
* Body Mass Index in the range of 18-30
* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any regular medications (except the contraceptive pill)

Exclusion Criteria:

* Currently any regular medications (except the contraceptive pill)
* History or current significant psychiatric illness
* Current alcohol or substance misuse disorder
* History or current significant hepatic disease
* History or current significant neurological condition (e.g. epilepsy)
* History of haemorrhagic stroke or lacunar infarct
* Known hyperglycaemia/pre-diabetes
* Known hypersensitivity to the study drug (i.e. simvastatin) or sucrose
* Pregnant, breast feeding, women of child-bearing potential not using appropriate contraceptive measures
* Participation in a study that uses the same or similar computer tasks as those used in the present study
* Participation in a study that involves the use of a medication within the last three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
FERT | Day 7 of drug/placebo administration
  The effects of simvastatin on emotional processing using the Facial Expression Recognition Task (FERT).
  FERT is a computer-based tasks of emotional processing using facial expressions of basic emotions (happiness, fear, anger, disgust, sadness, surprise) displayed on the screen and participants are asked to correctly classify them. Each emotion is presented at different intensity levels. Responses are made via a button-press. Accuracy and reaction times are measured.

SECONDARY OUTCOMES:
EMEM | Day 7 of drug/placebo administration
  The effects of simvastatin on Emotional Memory Task (EMEM) scores. Recall and recognition of affective words displayed earlier in the testing session are tested. Responses are made via a button-press. Accuracy and reaction times are measured.
ECAT | Day 7 of drug/placebo administration
  The effects of simvastatin on Emotional Categorisation Task (ECAT) scores. Disagreeable or agreeable personality descriptions are presented and participants are asked to indicate whether they would like or dislike to be described as each of these characteristics. Responses are made via a button-press. Accuracy and reaction times are measured.
EREC | Day 7 of drug/placebo administration
  The effects of simvastatin on Emotional Recall Task (EREC) scores. Participants are asked to write down as many of the words as they can remember from the previous task. Responses are made via pencil and paper. Accuracy is measured.
FDOT | Day 7 of drug/placebo administration
  The effects of simvastatin on Faces Dot-probe Task (FDOT) scores. Participants carry out a computer-based task of attentional vigilance to happy or fearful faces, recorded from participants' response latency to indicate the alignment of a dot-probe appearing in the place of one of the faces. Responses are made via button-press. Accuracy and reaction times are measured.
PILT | Day 7 of drug/placebo administration
  The effects of simvastatin on Probabilistic Instrumental Learning Task (PILT) scores.
  Participants have to learn which shapes are associated with wins and losses. Responses are made via button-press. Sensitivity to reward is measured.
AVLT | Day 7 of drug/placebo administration
  The effects of simvastatin on Auditory Verbal Learning Task (AVLT) scores. Accuracy of recall on the auditory verbal learning task.
CRP | Day 7 of drug/placebo administration
  The effects of simvastatin on C-reactive Protein (CRP) levels. Phlebotomy is performed to obtain a sample of CRP at baseline and at day 7 of drug/placebo administration. Changes in CRP levels are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Giorgi R, Quinton AMG, Waters S, Cowen PJ, Harmer CJ. An experimental medicine study of the effects of simvastatin on emotional processing, reward learning, verbal memory, and inflammation in healthy volunteers. Psychopharmacology (Berl). 2022 Aug;239(8):2635-2645. doi: 10.1007/s00213-022-06156-y. Epub 2022 May 5. PMID 35511258